CLINICAL TRIAL: NCT01965600
Title: A Phase 1, Randomized, Double Blind, Placebo Controlled, Multiple Dose, 2 Way Crossover Study To Evaluate The Safety And Pharmacodynamic Effects Of Pf 06282999 Using An Endotoxin (Lipopolysaccharide) Induced Inflammatory Response Model In Healthy Adult Subjects
Brief Title: A Study To Evaluate The Safety And Effects On The Body Of An Investigational Drug Using An Endotoxin-Induced Inflammatory Response Model
Acronym: POM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5211007; 2013-001528-20 (EudraCT Number)
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Endotoxin challenge
MeSH Terms: interventions — 2-(6-(5-chloro-2-methoxyphenyl)-4-oxo-2-thioxo-3,4-dihydropyrimidin-1(2H)-yl)acetamide; Endotoxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo; Other: LPS
- Cohort 2 (Experimental)
  Interventions: Drug: PF-06282999; Drug: Placebo; Other: LPS

INTERVENTIONS:
Drug: PF-06282999 — Tablet, 125 mg, TID, 3 days, 1 of 2 periods
  Arms: Cohort 1
Drug: Placebo — Tablet, 0 mg, TID, 3 days, 1 of 2 periods
  Arms: Cohort 1
Other: LPS — IV bolus, 4 ng/kg, 1 day, QD, 2 of 2 periods
  Other Names: Endotoxin
  Arms: Cohort 1
Drug: PF-06282999 — Tablet, 500 mg, BID, 3 days, 1 of 2 periods
  Arms: Cohort 2
Drug: Placebo — Tablet, 0 mg, BID, 3 days, 1 of 2 periods
  Arms: Cohort 2
Other: LPS — IV bolus, 4 ng/kg, 1 day, QD, 2 of 2 periods
  Other Names: Endotoxin
  Arms: Cohort 2

SUMMARY:
An endotoxin challenge will be administered to healthy subjects to induce production of inflammatory markers. An investigational drug or placebo will be administered prior to the endotoxin challenge to assess the effect of the investigational drug on the markers of inflammation. Safety and tolerability will also be assessed.

DETAILED DESCRIPTION:
The trial was terminated on 25 March 2015 due to safety concerns regarding the administration of endotoxin and because of the uncertain availability of future endotoxin lots.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women (non-childbearing potential) between the ages of 18-40 years.
* Body Mass Index (BMI) 18-30 kg/m2 and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* History or evidence of habitual use of tobacco- or nicotine-containing products within 3 months of screening.
* History of frequent headaches or migraines (>3 per month), or headaches from an absence of caffeine.
* Caffeine consumption in excess of 3 cups per day.
* Subjects who have experienced cold/flu symptoms (ie, runny nose, cough, and/or fever) within 2 weeks of the first administration of study drug/placebo of each period.
* History of recurrent or chronic infections of any type such as tuberculosis, sinusitis, urinary tract infection, respiratory tract or dental (abscess) infection, etc. Also excluded are subjects with recurrent oral or genital herpes, recurrent herpes zoster, or any infection otherwise judged by the investigator to have the potential for worsening if enrolled in this study.
* Treatment with LPS in the past 12 months and/or a history of an allergic type reaction or known hypersensitivity to endotoxin at any time.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - (Drug Shipment Address ONLY) Duke University Health Systems (DUHS) Investigational Drug Services, Durham, North Carolina
  - Duke Clinical Research Unit, Durham, North Carolina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5211007&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%20And%20Effects%20On%20The%20Body%20Of%20An%20Investigational%20Drug%20Using%20An%20Endotoxin-Induced%20Inflammatory%20Response%20Mod

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06282999 125 mg TID Followed by Placebo: Participants received PF-06282999 125 milligrams (mg) three times daily (TID) orally in tablet form from Days 1 to 3 (approximately 8am, 2pm, 8pm). On Day 3, participants received a dose of lipopolysaccharide (LPS) as an intravenous (IV) bolus at a dose of 4 nanogram (ng)/kilogram (kg) over 45-60 seconds (secs) 2 hours after the morning dose of PF-06282999. The final dose of PF-06282999 125 mg was administered on the evening of Day 3. After about 15 days of washout, participants returned for the second period where they received placebo in the same manner as active treatment before.
- Placebo Followed by PF-06282999 125 mg TID: Participants received placebo orally via tablets. Placebo matching PF-06282999 125 mg TID were administered on Days 1-3 at approximately 8am, 2pm, and 8pm. 2 hours after the morning dose on Day 3, LPS as IV bolus at a dose of 4 ng/kg over 45-60 secs was administered. The final dose of placebo was administered on the evening of Day 3. Following a washout of about 15 days, participants returned for the second period where they received PF-06282999 125 mg TID in the same manner as placebo in the first period.
- PF-06282999 500 mg BID Followed by Placebo: Participants received PF-06282999 500 milligrams (mg) twice daily (BID) orally in tablet form from Days 1 to 3 (8am and 8pm). On Day 3, participants received a dose of lipopolysaccharide (LPS) as an intravenous (IV) bolus at a dose of 4 ng/kg over 45-60 seconds (secs) 2 hours after the morning dose of PF-06282999. A final dose of PF-06282999 500 mg was administered on the evening of Day 3. After about 15 days of washout, participants returned for the second period where they received placebo in the same manner as active treatment before.
- Placebo Followed by PF-06282999 500 mg BID: Participants received placebo orally via tablets. Placebo matching PF-06282999 500 mg BID were administered on Days 1-3 at 8am and 8pm. 2 hours after the morning dose on Day 3, LPS as IV bolus at a dose of 4 ng/kg over 45-60 secs was administered. The final dose of placebo was administered on the evening of Day 3. Following a washout of about 15 days, participants returned for the second period where they received PF-06282999 500 mg BID in the same manner as placebo in the first period.
Period: First Intervention
Arm/Group | PF-06282999 125 mg TID Followed by Placebo | Placebo Followed by PF-06282999 125 mg TID | PF-06282999 500 mg BID Followed by Placebo | Placebo Followed by PF-06282999 500 mg BID
Started | 6 | 8 | 5 | 4
Received at Least One Dose of Drug | 6 | 8 | 5 | 4
Completed | 6 | 8 | 5 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of Approximately 15 Days
Arm/Group | PF-06282999 125 mg TID Followed by Placebo | Placebo Followed by PF-06282999 125 mg TID | PF-06282999 500 mg BID Followed by Placebo | Placebo Followed by PF-06282999 500 mg BID
Started | 6 | 8 | 5 | 4
Completed | 4 | 4 | 3 | 2
Not Completed | 2 | 4 | 2 | 2
Not completed — Study terminated by Sponsor | 1 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Did not meet entrance criteria | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Second Intervention
Arm/Group | PF-06282999 125 mg TID Followed by Placebo | Placebo Followed by PF-06282999 125 mg TID | PF-06282999 500 mg BID Followed by Placebo | Placebo Followed by PF-06282999 500 mg BID
Started | 4 | 4 | 3 | 2
Completed | 4 | 4 | 1 | 0
Not Completed | 0 | 0 | 2 | 2
Not completed — Study terminated by Sponsor | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All 23 participants who were randomized to study treatment and who received at least 1 dose of study drug were included in the baseline analysis.
Groups:
- All Participants: Participants received PF-06282999 125 mg TID or 500 mg BID or matching placebo orally in tablet form from Days 1 to 3. On Day 3, participants received a dose of LPS as an IV bolus at a dose of 4 ng/kg over 45-60 secs 2 hours after the morning dose of PF-06282999 or matching placebo. A final dose of PF-06282999 or matching placebo was administered on the evening of Day 3. Period 2 started after a washout period of approximately 15 days with at least 21 days in between administration of LPS. Participants who took active treatment (PF-06282999) in Period 1 received placebo in Period 2 and vice versa.
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Peak Myeloperoxidase (MPO) Activity Following Inflammatory Stimulus
Description: MPO is a heme-containing peroxidase enzyme produced in the bone marrow and stored in the azurophilic granules of neutrophils, where it constitutes up to 5% of the cellular protein. Since PF-06282999 is a mechanism-based inactivator of MPO, it is of interest to evaluate the level of MPO activity in order to investigate the inhibition activity of PF-06282999.
Time Frame: Days 1, 3-5
Population: Due to early termination of the study, there was not enough participants to perform meaningful analysis on this endpoint. As such, no analysis was done.
Groups:
- PF-06282999 125 mg TID: All participants who received PF-06282999 125 mg TID orally in tablet form from Days 1 to 3 (approximately 8am, 2pm, 8pm) in either Periods 1 or 2 are pooled in one group. On Day 3, participants received a dose of lipopolysaccharide (LPS) as an intravenous (IV) bolus at a dose of 4 nanogram (ng)/kilogram (kg) over 45-60 seconds (secs) 2 hours after the morning dose of PF-06282999. The final dose of PF-06282999 125 mg was administered on the evening of Day 3.
- Placebo: All participants who received placebo in either Periods 1 or 2 are pooled in 1 group. Placebo matching either PF-06282999 125 mg TID or 500 mg twice daily (BID) were administered on Days 1-3 of each period. 2 hours after the morning dose on Day 3, LPS as IV bolus at a dose of 4 ng/kg over 45-60 secs was administered. The final dose of placebo was administered on the evening of Day 3.
- PF-06282999 500 mg BID: All participants who received PF-06282999 500 mg BID orally in tablet form from Days 1 to 3 (8am and 8pm) in either Periods 1 or 2 are pooled in 1 group. On Day 3, participants received a dose of lipopolysaccharide (LPS) as an intravenous (IV) bolus at a dose of 4 ng/kg over 45-60 seconds (secs) 2 hours after the morning dose of PF-06282999. A final dose of PF-06282999 500 mg was administered on the evening of Day 3.
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: MPO Activity (Area Under the Concentration-time Profile From 0.5 to 2 Hours [AUC0.5-2hrs]) Following Inflammatory Stimulus
Description: as for outcome 1
Time Frame: Days 1, 3-5
Population: as for outcome 1
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: MPO Activity (Area Under the Concentration-time Profile From 0 to 2 Hours [AUC0-2hrs]) Following Inflammatory Stimulus
Description: as for outcome 1
Time Frame: Days 1, 3-5
Population: as for outcome 1
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Withdrawals Due to TEAEs
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as newly occurring AEs or those worsening after first dose. Due to early termination of the study, only AE data from partial enrollment are reflected and comparisons between treatment arms should not be attempted.
Time Frame: From Day 0 till approximately 7-10 days following the last dose of PF-06282999/Placebo in Period 2 (up to approximately 2 months)
Population: All participants who received at least 1 dose of study medication (including LPS) were included in the safety analyses and listings.
Measure: Number; unit: participants
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 10 | 19 | 7
participants
  Participants with TEAEs | 10 | 17 | 5
  Participants with SAEs | 0 | 0 | 0
  Participants discontinued permanently due to TEAEs | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, coagulation, liver function, renal function, electrolytes, clinical chemistry, and urinalysis (dipstick and microscopy). Due to early termination of the study, only laboratory data from partial enrollment are reflected and comparisons between treatment arms should not be attempted.
Time Frame: Baseline up to 7-10 days following the last dose of PF-06282999/Placebo in Period 2
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 10 | 19 | 7
participants | 5 | 8 | 5

6. Primary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Categorical Summarization Criteria
Description: Categorical summarization criteria in vital signs included: sitting, supine, and standing systolic blood pressure (SBP) of less than (<)90 millimeters of mercury (mm Hg) or change (increase [inc] or decrease [dec]) in sitting, supine and standing SBP of more than or equal to (>=)30 mm Hg; supine, sitting, and standing diastolic blood pressure (DBP) of <50 mm Hg or change (inc or dec) in sitting, supine, and standing DBP of >=20 mm Hg; supine and sitting pulse rate (PR) of <40 or more than (>)120 beats per minute (bpm); and standing PR of <40 or >140 bpm. Due to early termination of the study, only vital signs data from partial enrollment are reflected and comparisons between treatment arms should not be attempted.
Time Frame: Screening and Days 1-2, 4-5, and approximately 7-10 days following the last dose of PF-06282999/Placebo in Period 2 for orthostatic (orth) measurements; Day 3 for supine measurements
Population: All participants who received at least 1 dose of study medication (including LPS) were included in the safety analyses and listings. n=number of participants evaluable for that parameter
Measure: Number; unit: participants
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 10 | 19 | 7
participants
  Orthostatic SBP <90 mm Hg (n=0,1,0) | 0 | 0 | 0
  Orthostatic DBP <50 mm Hg (n=0,1,0) | 0 | 0 | 0
  Orthostatic PR <40 bpm (n=0,1,0) | 0 | 0 | 0
  Orthostatic supine SBP <90 mm Hg (n=10,18,7) | 0 | 0 | 0
  Orthostatic sitting SBP <90 mm Hg (n=1,0,0) | 0 | 0 | 0
  Orthostatic standing SBP <90 mm Hg (n=10,17,6) | 0 | 0 | 0
  Orthostatic supine DBP <50 mm Hg (n=10,18,7) | 0 | 0 | 0
  Orthostatic sitting DBP <50 mm Hg (n=1,0,0) | 0 | 0 | 0
  Orthostatic standing DBP <50 mm Hg (n=10,17,6) | 0 | 0 | 1
  Orthostatic supine PR <40 bpm (n=10,18,7) | 0 | 0 | 0
  Orthostatic supine PR >120 bpm (n=10,18,7) | 0 | 0 | 0
  Orthostatic sitting PR <40 bpm (n=1,0,0) | 0 | 0 | 0
  Orthostatic standing PR <40 bpm (n=10,17,6) | 0 | 0 | 0
  Orthostatic standing PR >140 bpm (n=10,17,6) | 0 | 0 | 0
  Supine SBP <90 mm Hg (n=10,17,5) | 0 | 2 | 0
  Supine DBP <50 mm Hg (n=10,17,5) | 1 | 2 | 1
  Supine PR <40 bpm (n=10,17,5) | 0 | 0 | 0
  Supine PR >120 bpm (n=10,17,5) | 1 | 4 | 0
  Increase in orth supine SBP >=30 mm Hg (n=10,18,7) | 1 | 0 | 0
  Inc in orth standing SBP >=30 mm Hg (n=10,17,6) | 0 | 0 | 0
  Inc in orth supine DBP >=20 mm Hg (n=10,18,7) | 0 | 0 | 0
  Inc in orth standing DBP >=20 mm Hg (n=10,17,6) | 0 | 0 | 0
  Inc in supine SBP >=30 mm Hg (n=10,17,5) | 0 | 4 | 1
  Inc in supine DBP >=20 mm Hg (n=10,17,5) | 1 | 3 | 0
  Dec in orth supine SBP >=30 mm Hg (n=10,18,7) | 0 | 1 | 0
  Dec in orth standing SBP >=30 mm Hg (n=10,17,6) | 0 | 2 | 0
  Dec in orth supine DBP >=20 mm Hg (n=10,18,7) | 1 | 0 | 1
  Dec in orth standing DBP >=20 mm Hg (n=10,17,6) | 0 | 1 | 1
  Dec in supine SBP >=30 mm Hg (n=10,17,5) | 1 | 1 | 1
  Dec in supine DBP >=20 mm Hg (n=10,17,5) | 1 | 4 | 2

7. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Values Meeting Categorical Summarization Criteria
Description: Criteria for ECG (12-lead) values meeting categorical summarization criteria were: the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval >=300 milliseconds (msec) and increase from baseline >=25/50%; time from the beginning of the ECG Q wave to the end of the S wave corresponding to ventricular depolarization (QRS) interval >=140 msec and increase of >=50%; the beginning of the Q wave to the end of the T wave corresponding to electrical systole (QT) interval >=500 msec; QT corrected using the Fridericia formula (QTcF) of 450 to <480 msec, 480 to <500 msec, and >=500 msec, or an increase of 30 to <60 msec or >=60 msec. Due to early termination of the study, only ECG data from partial enrollment are reflected and comparisons between treatment arms should not be attempted.
Time Frame: Screening; Days 1-5 and approximately 7-10 days following the last dose of PF-06282999/Placebo in Period 2
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 10 | 19 | 7
participants
  PR interval >=300 msec | 0 | 0 | 0
  QRS >=140 msec | 0 | 0 | 0
  QT >=500 msec | 0 | 0 | 0
  QTcF 450 to <480 msec | 0 | 2 | 0
  QTcF 480 to <500 msec | 0 | 0 | 0
  QTcF >=500 msec | 0 | 2 | 0
  PR interval increase >=25/50% | 0 | 0 | 0
  QRS increase >=50% | 0 | 0 | 0
  QTcF increase 30 to <60 msec | 0 | 3 | 1
  QTcF increase >=60 msec | 1 | 2 | 0

8. Primary Outcome: Number of Participants With Abnormal Urinary Biomarker Values
Description: Urinary biomarkers included albumin, neutrophil gelatinase-associated lipocalin (NGAL) and Cystatin-C.
Time Frame: Days 1-3 prior to dosing with PF-06282999/Placebo; and Days 4-5
Population: Analysis not done due to early termination of study.
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Concentrations of TNF-alpha, IL-1 Beta, IL-6, IL-8, and hsCRP
Description: The effect of multiple oral doses of PF-06282999 on inflammatory biomarkers was a secondary objective in this study. The biomarkers are tumor necrosis factor (TNF)-alpha, interleukin (IL)-1 beta, IL-6, IL-8, and high-sensitivity C-reactive protein (hsCRP).
Time Frame: Days 1, 3, and 4
Population: as for outcome 1
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Peak (AUC0.5-2hours and AUC0-2hours) of MPO Activity/MPO Mass
Description: as for outcome 1
Time Frame: Days 1, 3-5
Population: as for outcome 1
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-06282999
Time Frame: Day 3
Population: as for outcome 1
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Area Under the Concentration-time Profile From Time 0 to End of Dosing Interval, Tau (AUCtau) of PF-06282999
Time Frame: Day 3
Population: Due to early termination of the study, no data was collected for this endpoint.
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Time to Cmax (Tmax) of PF-06282999
Time Frame: Day 3
Population: Due to early termination of the study, no data was collected for this endpoint.
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through and including 28 calendar days after the last administration of the investigational product, up to approximately 2 months.
Description: All treated participants were analyzed for AEs. The same event may appear as both an AE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-06282999 125 mg TID | Placebo | PF-06282999 500 mg BID
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/19 | 0/7
Other Adverse Events (participants affected / at risk) | 10/10 | 17/19 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06282999 125 mg TID (N=10) | Placebo (N=19) | PF-06282999 500 mg BID (N=7)
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 7 | 13 | 4
Eye pain (Eye disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2
Chills (General disorders) | 8 | 11 | 3
Fatigue (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 10 | 13 | 3
Body temperature increased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 9 | 3
Headache (Nervous system disorders) | 8 | 13 | 4
Lethargy (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 3 | 1
Pallor (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to early study termination, PK, PD, or biomarker changes assessments were incomplete and there was only safety data from partial enrollment. As such, it was not possible to have meaningful interpretation and/or comparison of these data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.